CLINICAL TRIAL: NCT04673474
Title: A PhaseⅠFood-Effect Study of Hemay022 in Healthy Subjects
Brief Title: A Food-Effect Study of Hemay022 in Healthy Participants
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Hemay Oncology Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HM022BC1S02
Record Dates: First submitted 2020-12-09; First posted 2020-12-17 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2020-12

CONDITIONS: Food-drug Interaction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Hemay022 Period 1, Fasted control → Period 2, Fed control
  Interventions: Drug: Hemay022
- Arm B (Experimental): Hemay022 Period 1, Fed control → Period 2, Fasted control
  Interventions: Drug: Hemay022

INTERVENTIONS:
Drug: Hemay022 — Participants will receive a single oral dose of Hemay022 tablet in fasted condition on Day 1 of treatment period 1 followed by a single oral dose of Hemay022 tablet in fed condition on Day 8 of treatment period 2. A washout period of 7 days will be maintained between the 2 treatment periods.
  Arms: Arm A
Drug: Hemay022 — Participants will receive a single oral dose of Hemay022 tablet in fed condition on Day 1 of treatment period 1 followed by a single oral dose of Hemay022 tablet in fasted condition on Day 8 of treatment period 2. A washout period of 7 days will be maintained between the 2 treatment periods.
  Arms: Arm B

SUMMARY:
The primary objective of this study is to determine the effect of food in healthy participants on the bioavailability of Hemay022 following single dose administration with and without a meal.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-40 years old, the ratio of male to female is 1:1, the age difference of the same batch of subjects is less than 10 years;
2. Weight: male should not be less than 50kg, female should be no less than 45kg, body mass index (BMI) [=weight (kg)/height 2 (m2)] between 19-24 (including boundary values);
3. 90mmHg≤systolic blood pressure≤140mmHg, 60mmHg≤diastolic blood pressure≤90 mmHg, 55 beats/min≤pulse≤100 beats/min, 12 breaths/min≤respiration≤24 breaths/min, normal body temperature;
4. Before the trial, the subjects have understood the nature, significance, possible benefits and possible inconveniences and potential dangers of the trial in detail, and volunteered to participate in the clinical trial, can communicate well with the investigator, comply with the requirements of the entire study, and Signed a written informed consent form.

Exclusion Criteria:

1. Participated in other drug clinical trials within 3 months;
2. (Inquiry)Diseases with abnormal clinical manifestations that need to be excluded, including but not limited to diseases of the nervous system, cardiovascular system, blood and lymphatic system, immune system, kidney, liver, gastrointestinal tract, respiratory system, metabolism and bones;
3. (Inquiry)Those who have a history of severe vomiting, diarrhea or any other diseases or physiological conditions that can interfere with the study results within 7 days before the trial;
4. (Inquiry)People with a history of specific allergies (asthma, urticaria, eczema, etc.), or allergies (such as those who are allergic to two or more drugs, food or pollen), or those who are known to be allergic to tiniba drugs;
5. (Inquiry) Those who lost blood or donated more than 400ml of blood within 3 months before this clinical trial, or plan to donate blood during the trial;
6. Inquiry) Pregnant or lactating female, or subjects (including male subjects) have a childbirth plan or sperm donation plan within 3 months after the last dose, unwilling or unwilling Those who take effective contraceptive measures;
7. General physical examination and laboratory examination (blood routine, stool routine, blood biochemistry, coagulation function, urine routine, blood human chorionic gonadotropin/urinary pregnancy (female), etc.) within 7 days before the test, 6 months before the test The result of internal chest radiograph is judged by clinicians as abnormal and clinically significant;
8. Subjects whose left ventricular ejection fraction (LVEF) measured by MUGA scan or echocardiography is less than 50%;
9. Patients with clinically significant ECG abnormalities in the 14 days before the test, including: QTc (corrected by bazett or fridericia) interval prolonged (≥450ms) on the screening ECG, QRS>120ms;
10. One or more test results of hepatitis B surface antigen, hepatitis C virus antibody, anti-human immunodeficiency virus antibody or Treponema pallidum antibody are positive;
11. (Inquiry) Those who have suffered from a clinically significant disease or have undergone major surgery within 3 months before the trial;
12. (Inquiry) Drinking more than 14 units per week (1 unit = 17.7 mL ethanol, ie 1 unit = 357 mL of beer with 5% alcohol content or 43 mL of liquor with 40% alcohol content or 147 mL of wine with 12% alcohol content), or those who cannot abstain from alcohol during the test;
13. (Inquiry) Those who smoked more than 5 cigarettes a day on average in the 3 months before the test, or who could not stop using any tobacco products during the test;
14. (Inquiry) People who drank excessive amounts of tea, coffee and/or caffeine-rich beverages (more than 8 cups, 1 cup = 250 mL) during the 3 months before screening;
15. (Inquiry) Have taken grapefruit (including grapefruit), pomegranate, lime, carambola, dragon fruit, mango and other fruits or food or beverages prepared therefrom within 7 days before screening;
16. (Inquiry) People who have eaten chocolate, caffeine-rich, xanthine-rich food or beverages and other special diets that affect drug absorption, distribution, metabolism, and excretion during the period from screening to -1 day;
17. (Inquiry) Those who cannot eat or have difficulty swallowing, have special dietary requirements and/or cannot follow a unified diet;
18. (Inquiry) Those who have a history of asthma or seizures;
19. (Inquiry) Those who have used any drugs within 1 month before the trial;
20. (Inquiries) Machine operators who are engaged in high-altitude operations, motor vehicle driving and other dangerous machinery operators;
21. (Inquiry) Those who cannot tolerate venipuncture and/or have a history of fainting blood and needles;
22. (Inquiry) People with a history of hereditary galactose intolerance, lactase deficiency or glucose-galactose malabsorption;
23. (Inquiry) Those who have used any drugs within one year before the trial;
24. Alcohol breath test results greater than 0.0mg/100ml or those who are positive for drug abuse screening (morphine, methamphetamine, ketamine, amphetamine, tetrahydrocannabinol acid, cocaine) );
25. Subjects considered by the investigator to have poor compliance or have any factors that are not suitable for participating in this trial.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-12-09 (Actual); Primary Completion 2021-02-04 (Actual); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Cmax | Day 1: 0-48 hours; Day 8: 0-48 hours
  Maximum Observed Plasma Concentration for Hemay022
Tmax | Day 1: 0-48 hours; Day 8: 0-48 hours
  Time to Reach the Maximum Observed Plasma Concentration (Cmax) for Hemay022
AUC0-t | Day 1: 0-48 hours; Day 8: 0-48 hours
  AUC 0-t: Area Under the Concentration-time Curve From Zero (Pre-dose) to Time of Last Quantifiable Concentration for Hemay022
AUC0-∞ | Day 1: 0-48 hours; Day 8: 0-48 hours
  Area Under the Plasma Concentration-time Curve from Time 0 to Infinite Time for Hemay022

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, China